CLINICAL TRIAL: NCT06592612
Title: Second-line Systemic Therapy with or Without Stereotactic Body Radiotherapy (SBRT) for Oligoprogressive Hepatocellular Carcinoma After Standard First-line Systemic Treatment: a Prospective, Randomized, Phase II Study
Brief Title: Second-line Systemic Therapy Combined with SBRT for HCC with Oligoprogression After Standard First-line Systemic Treatment
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Chen Min-Shan, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B2024-428-01
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hepatocellular Carcinoma; Oligoprogression
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Arm (Active Comparator): Patients in the control arm will receive second-line systemic therapy until disease progression is confirmed by imaging or until they are unable to continue systemic therapy due to adverse events. The following stipulations apply to the second-line treatment drugs: for patients who received bevacizumab combined with atezolizumab/sintilimab as the first-line treatment, lenvatinib or regorafenib will be used for second-line treatment; for patients who received lenvatinib with or without PD-1 antibody as the first-line treatment, regorafenib combined with another PD-1 antibody will be used for second-line treatment.
  Interventions: Drug: Second-line systemic therapy
- SBRT Arm (Experimental): Patients in the SBRT arm will also receive second-line systemic therapy until disease progression is confirmed by imaging or until they are unable to continue systemic therapy due to adverse events. The choice and stipulations for second-line systemic therapy drugs are the same as those for the control arm. SBRT will be administered to all oligoprogressive lesions and must begin within 2 weeks after the start of second-line therapy. Systemic therapy will not be paused during SBRT. Patients who do not withdraw from the study will not receive crossover treatment; however, if a patient in the control group withdraws from the study due to tumor progression and is assessed as suitable for SBRT, salvage SBRT will be administered promptly.
  Interventions: Radiation: SBRT and second-line systemic therapy

INTERVENTIONS:
Radiation: SBRT and second-line systemic therapy — Patients in the SBRT arm will receive second-line systemic therapy combined with SBRT. The choice and stipulations for second-line systemic therapy drugs are the same as those for the control arm.SBRT will be administered to all oligoprogressive lesions and must begin within 2 weeks after the start of second-line therapy. Systemic therapy will not be paused during SBRT. Patients who do not withdraw from the study will not receive crossover treatment; however, if a patient in the control group withdraws from the study due to tumor progression and is assessed as suitable for SBRT, salvage SBRT will be administered promptly.
  Arms: SBRT Arm
Drug: Second-line systemic therapy — Patients in the control arm will receive second-line systemic therapy. The following stipulations apply to the second-line treatment drugs: for patients who received bevacizumab combined with atezolizumab/sintilimab as the first-line treatment, lenvatinib or regorafenib will be used for second-line treatment; for patients who received lenvatinib with or without PD-1 antibody as the first-line treatment, regorafenib combined with another PD-1 antibody will be used for second-line treatment.
  Arms: Control Arm

SUMMARY:
Approximately 70% of hepatocellular carcinoma (HCC) patients are diagnosed at an advanced stage, with no opportunity for curative treatments. For these patients, systemic therapies are the main treatment modalities. However, the objective response rates of first-line systemic treatments are currently only 20-35%, and most patients inevitably develop drug resistance and disease progression during treatment, thus taking second-line therapies. Second-line treatment options include regorafenib, pembrolizumab, and others, but clinical studies have shown a median progression-free survival of only 2.6-3.1 months, indicating an urgent need to improve efficacy.

Stereotactic body radiotherapy (SBRT) has been widely used in recent years for curative treatment of early-stage liver cancer or as neoadjuvant and adjuvant therapy for patients with portal vein tumor thrombus. It is one of the important approaches in the multidisciplinary management of HCC. Researches have shown that SBRT has a synergistic effect with systemic drug therapy, potentially enhancing the efficacy of targeted and immunotherapies. Therefore, this study aims to conduct a prospective, randomized, controlled phase II clinical trial in patients with oligoprogressive HCC after standard first-line systemic treatment to evaluate whether adding SBRT to second-line systemic therapy can improve the efficacy of second-line treatment. The primary endpoint of the study is progression-free survival (PFS), while secondary endpoints include overall survival (OS), objective response rate (ORR), and treatment-related adverse events. We aim to comprehensively assess the effectiveness and safety of combining SBRT with second-line systemic therapy in treating oligoprogressive HCC patients.

ELIGIBILITY:
Inclusion Criteria:

1. KPS (Karnofsky Performance Status) score ≥ 80;
2. Pathologically, or clinically diagnosed hepatocellular carcinoma (HCC) based on the " Chinese Guidelines for the Diagnosis and Treatment of Hepatocellular Carcinoma (2024 Edition) ";
3. Patients with oligoprogression after first-line standard systemic therapy (bevacizumab combined with atezolizumab/sintilimab or lenvatinib with or without PD-1 antibody).

   Definition of oligoprogression: 1-5 progressive lesions involving 1-3 organs/systems, including: (1)The maximum diameter of a target lesion, as assessed by RECIST 1.1 criteria, increases by more than 20% compared to baseline, with an absolute increase of >5 mm; (2) The maximum diameter of a target lesion increases by more than 20% compared to baseline on two consecutive evaluations (at least 2 months apart), regardless of whether the absolute increase is >5 mm; (3) The appearance of a new intrahepatic lesion ≥1 cm with typical imaging characteristics of HCC; 4) The appearance of any new extrahepatic lesion or bone metastasis, regardless of size; 5) Any new FDG-avid lesion confirmed by PET/CT, or an increase in SUVmax of more than 30% with an absolute increase of >0.8 SUV; 6) In the case of lymph node metastasis, each lymphatic drainage area is counted as one organ.
4. All oligoprogressive lesions are deemed suitable for radiotherapy, with a maximum diameter of any single oligoprogressive lesion not exceeding 5 cm, and at least one measurable lesion (according to RECIST v1.1 criteria); bone metastases without soft tissue formation are eligible but considered non-measurable lesions; if bone metastases have soft tissue formation and meet measurable criteria, they are considered measurable lesions;
5. Child-Pugh score for liver function ≤ 7;
6. Estimated life expectancy greater than 3 months;
7. Function of essential organs meets the following criteria: white blood cells ≥ 3.0 × 10^9/L, neutrophils ≥ 1.5 × 10^9/L, platelets ≥ 50.0 × 10^9/L, hemoglobin ≥ 90 g/L; serum albumin ≥ 2.8 g/dL; total bilirubin ≤ 1.5 × ULN, ALT/AST/ALP ≤ 2.5 × ULN; serum creatinine ≤ 1.5 × ULN or creatinine clearance > 60 mL/min; no severe organic disease;
8. Participants must have the ability to understand and voluntarily sign a written informed consent form. Consent must be obtained before any specific study procedures begin, and the participant must agree to follow the medication and post-operative follow-up requirements outlined in the study design.

Exclusion Criteria:

1. Received first-line treatment other than bevacizumab combined with atezolizumab/sintilimab or lenvatinib with or without PD-1 antibody;
2. Tumor progression within 3 months after first-line standard systemic therapy;
3. Experienced ≥ Grade 3 severe adverse reactions after first-line standard therapy;
4. Brain metastasis with hemorrhage at baseline or after first-line systemic therapy;
5. Previous radiotherapy to the site of the oligoprogressive lesion;
6. Active bleeding (e.g., hematemesis, hemoptysis) within 2 months before enrollment;
7. Received any other antitumor drug therapy or local treatment within 3 months before enrollment;
8. Severe impairment of the heart, lungs, kidneys, or other vital organs, active infections (other than viral hepatitis), or other severe comorbidities that make the patient unable to tolerate treatment;
9. History of other malignancies, except for non-melanoma skin cancer, carcinoma in situ of the cervix, or early-stage prostate cancer that has been cured;
10. Presence of autoimmune diseases or other conditions requiring long-term use of steroids;
11. Known or suspected allergy to the study drugs or any drugs related to this trial;
12. History of organ transplantation;
13. Pregnant or breastfeeding women;
14. Other factors that may affect the patient's enrollment and assessment results;
15. Refusal to follow the follow-up requirements set by this study protocol or refusal to sign the informed consent form.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
progression-free survival, PFS | From date of treatment beginning until the date of follow-up completion, up to 2 year.
  PFS is defined as the time from treatment to the first confirmed disease progression based on imaging assessment according to the RECIST v1.1 criteria.

SECONDARY OUTCOMES:
objective response rate，ORR | From date of treatment beginning until the date of follow-up completion, up to 2 year.
  The ratio of patients achieving the best efficacy of the corresponding interventions, including complete response (CR) and partial response (PR), to all patients in the arm.
overall survival, OS | From date of treatment beginning until the date of follow-up completion, up to 2 year.
  OS is defined as the time from treatment beginningto death from any cause
Incidence of adverse events (safety ) | From date of treatment beginning until the date of follow-up completion, up to 2 year.
  Treatment-related adverse events are evaluated according to the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (CTCAE 5.0)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP